CLINICAL TRIAL: NCT00263939
Title: A Randomized Trial of Home Self-Efficacy Enhancement
Brief Title: Homing in on Health: Study of a Home Delivered Chronic Disease Self Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Anthony Jerant, MD, University of California Davis School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01HS013603 (AHRQ)
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes Mellitus; Congestive Heart Failure; Arthritis; COPD; Depression
Keywords: chronic disease; patient education; self-efficacy; self-management
MeSH Terms: conditions — Diabetes Mellitus; Heart Failure; Arthritis; Pulmonary Disease, Chronic Obstructive; Depression; Chronic Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 - In home intervention (Experimental): In home (face to face) delivery of the study intervention, Homing in on Health
  Interventions: Behavioral: Homing in on Health
- 2 - Telephone intervention (Experimental): Telephone delivery of the study intervention, Homing in on Health
  Interventions: Behavioral: Homing in on Health
- 3 - Usual care (No Intervention): Patients receiving the care their usual health providers supply, without an study intervention

INTERVENTIONS:
Behavioral: Homing in on Health — A peer (non-health professional) delivered intervention to enhance patient self-efficacy for chronic disease self-management. Developed as a modification of the Stanford Chronic Disease Self-Management Program.
  Arms: 1 - In home intervention; 2 - Telephone intervention

SUMMARY:
The purpose of the study is to determine the effectiveness of a home-delivered variant of the chronic disease self management program in improving health outcomes in patients with chronic conditions.

DETAILED DESCRIPTION:
Key reasons for the "quality chasm" between current and ideal chronic illness care are that our health care system is insensitive to patient preference, provider-driven, and disease-focused. By contrast, a common goal among proposed patient-centered care models is to foster continuous healing relationships between patients and the health care system. Such relationships allow patients to receive care over time via a variety of communication media, rather than just via periodic office visits. Home health care can foster such relationships and improve outcomes for patients with a variety of conditions. Home interventions may be particularly useful in caring for the growing number of people with chronic illnesses accompanied by functional limitations that reduce their access to community-based interventions such as group self-care classes. However, trials comparing the effectiveness of the wide array of home care models are limited, and the mechanisms that underlie their effectiveness remain unclear.

This randomized controlled trial (RCT) of 3 groups, comparing the effectiveness and cost-effectiveness of 2 different home-based care models and usual care in improving chronic illness outcomes, will address these research gaps. The primary outcome will be health-related quality of life (HRQoL). We will also explore the mechanisms of effectiveness of home care through its influence on self-efficacy - beliefs patients have about their ability to successfully execute the actions required to achieve valued health outcomes - and adherence. The chronic illnesses targeted will be diabetes mellitus (DM), congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD), asthma, arthritis, and depression. The home care delivery media in the models will be in-person visits, and standard telephone calls. The study hypotheses are: a) Each of the 3 different home interventions will result in improvements in patient self-efficacy, adherence to care, and HRQoL compared with usual care but will not differ statistically; b) From the payer's perspective, all the interventions will be cost saving compared with usual care, and a standard telephone intervention will be the most cost saving; and c) Self-efficacy will improve temporally before adherence to care and HRQoL.

The research proven framework for improving patient self-efficacy that we will employ in our interventions, the Chronic Disease Self-Management Program (CDSMP), was developed at Stanford University. It was designed to be delivered by trained laypersons to groups of patients in community settings. The CDSMP developers will serve as consultants on our study, assisting us with modifying the program for delivery by trained lay visitors to individual patients in their homes.

ELIGIBILITY:
Inclusion Criteria:

* receive primary care 1 of 12 UC Davis Primary Care Network (PCN) offices
* live in a private home
* age 40 or older
* able to read and speak english
* Adequate vision and hearing to read study materials and use a standard telephone
* have one or more of the following conditions: arthritis, asthma, COPD, CHF, depression, DM
* suffer functional impairment as manifest by at least one of the following: self-reported impairment in at least 1 basic activity of daily living on Health Assessment Questionnaire (HAQ); or score higher than 3 on the 10-item version of the Center for Epidemiologic Studies Depression Scale (CES-D)

Exclusion criteria: see above

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2004-07; Primary Completion 2006-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Health related quality of life (HRQoL) at 2wks and 4wks during the intervention, immediately post intervention and at 6 months and 1 year post intervention

SECONDARY OUTCOMES:
self-care self-efficacy at 2wks and 4wks during the intervention, immediately post intervention and at 6 months and 1 year post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Jerant, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Jerant AF, von Friederichs-Fitzwater MM, Moore M. Patients' perceived barriers to active self-management of chronic conditions. Patient Educ Couns. 2005 Jun;57(3):300-7. doi: 10.1016/j.pec.2004.08.004. PMID 15893212
- [Background] Jerant A, DiMatteo R, Arnsten J, Moore-Hill M, Franks P. Self-report adherence measures in chronic illness: retest reliability and predictive validity. Med Care. 2008 Nov;46(11):1134-9. doi: 10.1097/MLR.0b013e31817924e4. PMID 18953223
- [Background] Jerant A, Chapman BP, Franks P. Personality and EQ-5D scores among individuals with chronic conditions. Qual Life Res. 2008 Nov;17(9):1195-204. doi: 10.1007/s11136-008-9401-y. Epub 2008 Oct 7. PMID 18839336
- [Result] Franks P, Chapman B, Duberstein P, Jerant A. Five factor model personality factors moderated the effects of an intervention to enhance chronic disease management self-efficacy. Br J Health Psychol. 2009 Sep;14(Pt 3):473-87. doi: 10.1348/135910708X360700. Epub 2008 Sep 20. PMID 18808733
- [Result] Jerant A, Moore M, Lorig K, Franks P. Perceived control moderated the self-efficacy-enhancing effects of a chronic illness self-management intervention. Chronic Illn. 2008 Sep;4(3):173-82. doi: 10.1177/1742395308089057. PMID 18796506
- [Result] Jerant A, Kravitz R, Moore-Hill M, Franks P. Depressive symptoms moderated the effect of chronic illness self-management training on self-efficacy. Med Care. 2008 May;46(5):523-31. doi: 10.1097/MLR.0b013e31815f53a4. PMID 18438201
- [Derived] Chapman BP, Franks P, Duberstein PR, Jerant A. Differences between individual and societal health state valuations: any link with personality? Med Care. 2009 Aug;47(8):902-7. doi: 10.1097/MLR.0b013e3181a8112e. PMID 19543121
- [Derived] Jerant A, Chapman BP, Duberstein P, Franks P. Is personality a key predictor of missing study data? An analysis from a randomized controlled trial. Ann Fam Med. 2009 Mar-Apr;7(2):148-56. doi: 10.1370/afm.920. PMID 19273870